CLINICAL TRIAL: NCT05177042
Title: A Phase 1b Open-Label, Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of ARV-110 in Combination With Abiraterone in Patients With Metastatic Prostate Cancer
Brief Title: Trial of ARV-110 and Abiraterone in Patients With Metastatic Castration Resistant Prostate Cancer (mCRPC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arvinas Androgen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Organization: Arvinas Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARV-110-mCRPC-103
Record Dates: First submitted 2021-11-19; First posted 2022-01-04 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer Metastatic
Keywords: Metastatic Prostate Cancer; Prostate Cancer; Castrate-Resistant; mCRPC; bavdegalutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral tablet(s) in combination with abiraterone and a corticosteroid. (Experimental): ARV-110 oral tablets in combination with abiraterone and a corticosteroid administered daily in 28 day cycles.
  Interventions: Drug: ARV-110 in Combination with Abiraterone

INTERVENTIONS:
Drug: ARV-110 in Combination with Abiraterone — ARV-110 oral tablets in combination with abiraterone and a corticosteroid administered daily in 28 day cycles

SUMMARY:
Phase 1b study to assess the combination of ARV-110 and abiraterone in patients with metastatic prostate cancer with rising PSA values on abiraterone.

ELIGIBILITY:
Inclusion Criteria:

1. Histological, pathological, or cytological confirmed diagnosis of adenocarcinoma of the prostate.
2. Ongoing treatment with stable doses of abiraterone (on an empty stomach) and a concomitant corticosteroid for metastatic castration-resistant prostate cancer (mCRPC) or for metastatic castration sensitive prostate cancer (mCSPC) until Cycle 1, Day 1 (C1D1).
3. Recent PSA values must demonstrate:

   1. Rising PSAs at least 16 weeks after initiation of abiraterone
   2. At least 2 PSA values that are higher than the PSA nadir on abiraterone, measured at a minimum of 1 week apart . The screening PSA for this study may be used as the 2nd PSA value.
4. No known radiographic evidence of disease progression while receiving abiraterone and clinically benefitting at the time of consent. If there is radiographic disease progression during screening, the patient may be considered eligible if, in the judgement of the investigator, the patient is clinically benefitting from abiraterone.
5. Ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) analogue or inhibitor, or orchiectomy (surgical or medical castration).
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

1. Previously treated with enzalutamide, apalutamide, darolutamide or experimental therapies (e.g., protein degraders or inhibitors) directed at the AR.
2. Treatment with any chemotherapy, investigational agents, immunotherapy, or hormonal therapy other than GnRH agonists within 28 days of the start of treatment on protocol.
3. Radiation therapy within 4 weeks of first dose of study drug or prior irradiation to >25% of the bone marrow.
4. Patients taking agents that are either a) sensitive P-glycoprotein (P-gp), breast cancer resistance protein (BCRP) substrates, or CYP3A4 substrates, b) P-gp, BCRP, CYP3A4, or CYP2D6 substrates that have a narrow therapeutic index, c) strong CYP3A4 inhibitors or inducers, or d) any other prohibited and/or restricted medications described in the protocol.
5. Major surgery (as judged by the Investigator) within 4 weeks of first dose of study drug.
6. Untreated brain metastases or brain metastases requiring steroids
7. Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
8. Any of the following in the previous 12 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association class II, III or IV), cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism, or other clinically significant episode of thromboembolic disease.
9. Any of the following in the previous 6 months: congenital long QT syndrome, Torsade de Pointes, arrhythmias (including sustained ventricular tachyarrhythmia and ventricular fibrillation), left anterior hemiblock (bifascicular block), or ongoing cardiac dysrhythmias of National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Grade ≥2, atrial fibrillation of any grade (Grade ≥2 in the case of asymptomatic lone atrial fibrillation)..
10. Hypertension that cannot be controlled by medications (>150/90 mmHg despite optimal medical therapy).
11. Active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus, hepatitis C virus, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
12. Active inflammatory gastrointestinal disease, uncontrolled chronic diarrhea, known diverticular disease, or previous gastric resection or lap band surgery. Gastroesophageal reflux disease is allowed except for if under treatment with proton pump inhibitors.
13. Patients with Child Pugh C.
14. Patients with electrolyte imbalances of hypokalemia, hypomagnesemia, and/or hypocalcemia.
15. Patients with QTcF ≥470 msec.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities of ARV-110 in combination with abiraterone | 4 weeks
  Dose limiting toxicities in first 4 weeks of the study combination treatment characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), timing, seriousness, and relationship to study drug
Number of Patients with Adverse Events as a measure of safety and tolerability of ARV-110 in combination with abiraterone | 35 days after subject discontinues study treatment
  Adverse events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug combination
Incidence of laboratory abnormalities as a measure of safety and tolerability of ARV-110 in combination with abiraterone | 35 days after subject discontinues study treatment
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), and timing.
Recommended Phase 2 dose (RP2D)/schedule for the combination | 4 weeks
  Dose limiting toxicities in first 4 weeks of the study combination treatment will be assessed to determine the dose of ARV-110 and abiraterone associated with acceptable safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (9):
  - Clinical Trial Site, Santa Monica, California
  - Clinical Trial Site, New Haven, Connecticut
  - Clinical Trial Site, Fort Myers, Florida
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Myrtle Beach, South Carolina
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Charlottesville, Virginia
- Canada (3):
  - Clinical Trial Site, Vancouver, British Columbia
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Montreal, Quebec
- France (3):
  - Clinical Trial Site, Caen, France
  - Clinical Trial Site, Paris, France
  - Clinical Trial Site, Villejuif, France
- United Kingdom (3):
  - Clinical Trial Site, London, England
  - Clinical Trial Site, Cardiff, Wales
  - Clinical Trial Site, Preston

IPD SHARING:
Plan to Share IPD: No